CLINICAL TRIAL: NCT03435016
Title: A Comparative Study of Magnetic Resonance Imaging, Ultrasound and Capsule Endoscopy of the Small and Large Intestine for Assessing Treatment Response in Known Crohn's Disease
Brief Title: A Comparative Study of MRI, US and CE for Assessing Treatment Response in Known Crohn's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sygehus Lillebaelt (Other)
Collaborators: Odense University Hospital (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Responsible Party: Principal Investigator, Michael Dam Jensen, Principal investigator, Sygehus Lillebaelt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ANDI-2
Record Dates: First submitted 2018-02-02; First posted 2018-02-15 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Ultrasonography; Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnosis (Other)
  Interventions: Diagnostic Test: Diagnostic work-up

INTERVENTIONS:
Diagnostic Test: Diagnostic work-up — Patients are examined with all modalities. MR enterocolonography, ultrasound, and small bowel capsule endoscopy are compared against ileocolonoscopy (gold standard).
  Other Names: Ileocolonoscopy; MR enterocolonography; Ultrasound; Small bowel colon capsule endoscopy

SUMMARY:
The aim of this study is to evaluate non-invasive imaging techniques for assessing treatment response in known Crohn's disease.

1. Comparing imaging modalities:

   The applicability of small bowel colon capsule endoscopy (SBCCE), magnetic resonance enterocolonography (MREC) and ultrasound (US) for diagnosing ulcer healing after medical treatment in patients with symptomatic Crohn's disease compared to ileocolonoscopy.
   1. Sensitivity and specificity for ulcer healing
   2. Changes in activity parameters for SBCCE, MREC and US before and after medical treatment.
   3. Feasibility of SBCCE, MREC and US for assessing treatment response in known Crohn's disease.
2. Treatment induced bowel wall alterations visualized with ultrasound:

   1. A non-blinded study of bowel wall changes detected with repeated US examination during medical treatment of known Crohn's disease.
   2. Changes in bowel wall thickness, vascularity and elastography parameters, and time to normalization of the bowel wall.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the applicability of SBCCE, MREC and US for diagnosing ulcer healing after medical treatment in patients with symptomatic CD compared to the current gold standard (ileocolonoscopy).

This is a prospective, blinded, multicenter study. Patients are recruited from 3 centers in the Region of Southern Denmark managing adult patients with inflammatory bowel diseases. Each patient goes through a standardized work-up including medical history, physical examination, C-reactive protein, fecal calprotectin, ileocolonoscopy, SBCCE, MREC and US before and 10-12 weeks after medical treatment with corticosteroids or biological therapy (Infliximab, Adalimumab, Vedolizumab or Ustekinumab). All examinations are reviewed and described in a standardized fashion. The radiologists and physicians describing SBCCE, MREC, and US are blinded to the findings at ileocolonoscopy and the other imaging modalities. Ileocolonoscopy serves as the diagnostic gold standard, and endoscopic disease activity is assessed with SES-CD.

LOGISTICS: Patients go through an accelerated diagnostic work-up at inclusion and after 10-12 weeks of medical treatment. In patients undergoing their first diagnostic work-up, ileocolonoscopy with biopsies is performed last to avoid false positive lesions at SBCCE. In patients with an established diagnosis, examinations can be performed in a random order provided that tissue samples are not taken during ileocolonoscopy. All diagnostic procedures should be completed within two weeks. If one imaging modality is contraindicated it is classified as "not performed". If ileocolonoscopy (gold standard) is contraindicated, the patient is excluded from the study. All radiological examinations are performed in the Department of Radiology, Lillebaelt Hospital Vejle. Ileocolonoscopy and SBCCE are performed at the local gastroenterology department.

During the pre- and post-treatment assessment, radiological examinations and SBCCE are analyzed by physicians blinded to the result of ileocolonoscopy and the other bowel examinations. However, at the post-treatment assessment, physicians are not blinded to the pre-treatment examinations. After completing all diagnostic procedures, the treating gastroenterologist is provided with the results of SBCCE, MREC and US.

EXTENDED ULTRASOUND STUDY: Patients are scheduled for additional US procedures after 2 and 4 weeks. Procedures are performed without blinding, i.e. the physician is aware of the results of the pre-treatment assessment and the preceding US examinations. If the bowel wall normalizes at week 2, the subsequent procedure is cancelled. Fecal calprotectin is measured before each US procedure.

ELIGIBILITY:
Inclusion Criteria:

* An established diagnosis of CD
* Age > 18 years
* Ileocolonoscopy: Endoscopically active CD (SES-CD ≥ 3)
* Clinically active CD (Harvey-Bradshaw Index ≥ 5 or Crohn's Disease Activity Index ≥ 150)
* Clinical indication for medical treatment with corticosteroids or biological therapy
* Signed informed consent

Exclusion Criteria:

* Acute bowel obstruction
* Intake of NSAIDs or acetylsalicylic acid ≤ 4 weeks before inclusion except prophylactic treatment with low dose Aspirin (≤ 150 mg per day)
* Pregnancy or lactation
* Alcohol or drug abuse
* Known gastrointestinal disorder other than inflammatory bowel disease
* Renal failure defined by a plasma-creatinine above the normal reference range
* Claustrophobia, cardiac pacemaker or implanted magnetic foreign bodies that precludes MREC
* Interpreter required or inability to understand the oral and written information
* Bowel surgery performed between pre- and post-treatment assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | 8-10 weeks
  Sensitivity and specificity of SBCCE, MREC and US for the diagnosis of ulcer healing in the terminal ileum and colon

SECONDARY OUTCOMES:
Diagnostic accuracy fCal | 8-10 weeks
  Sensitivity and specificity of fecal calprotectin for the diagnosis of ulcer healing in the terminal ileum and colon
Diagnostic accuracy CRP | 8-10 weeks
  Sensitivity and specificity of C-reactive protein for the diagnosis of ulcer healing in the terminal ileum and colon
Bowel wall thickening | 8-10 weeks
  Changes of bowel wall thickening (mm) assessed with US under medical treatment of Crohn's disease
Elastography | 8-10 weeks
  Changes of shear wave elastography (m/s) assessed with US under medical treatment of Crohn's disease
Ultrasound activity index | 8-10 weeks
  Changes of Limberg score assessed with US under medical treatment of Crohn's disease

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Jensen, MD, PhD, Principal Investigator — Lillebaelt Hospital Vejle
Locations (1):
- Sygehus Lillebaelt, Vejle, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will not be available to other researchers.

REFERENCES:
- [Derived] Brodersen JB, Rafaelsen SR, Nejatbakhsh E, Jensen MD. Assessment of transmural treatment response in known Crohn's disease: a prospective blinded study of the intermodality agreement between intestinal ultrasound and magnetic resonance enterography. BMJ Open Gastroenterol. 2026 Feb 9;13(1):e002175. doi: 10.1136/bmjgast-2025-002175. PMID 41663130